CLINICAL TRIAL: NCT06590909
Title: Fractional CO2 Laser for Delivery of Topical Insulin Versus Platelet Rich Plasma in Treatment of Atrophic Post Acne Scars: a Split Face Comparative Study
Brief Title: Fractional CO2 Laser Delivery of Topical Insulin Versus Platelet Rich Plasma in Treatment of Atrophic Post Acne Scars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Mohamed Gamal, principal investigator, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: treatment of post acne scars
Record Dates: First submitted 2024-06-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A prospective comparative split face study (Active Comparator)
  Interventions: Combination Product: Fractional CO2 laser assisted PDT

INTERVENTIONS:
Combination Product: Fractional CO2 laser assisted PDT — Comparative split face study: participants will be treated with fractional co2 laser on the whole face then applying topical insulin on the right side of the face and topical platelet rich plasma on the left side of the face.
  Other Names: topical platelet rich plasma

SUMMARY:
compare the efficacy and safety of treating atrophic post acne scars with topical insulin versus Platelet rich Plasma PRP combined with fractional ablative Co2 laser

DETAILED DESCRIPTION:
Acne vulgaris is a common cutaneous inflammatory disorder of the pilosebaceous unit, which runs a chronic course. The condition commonly manifests with papules, pustules, or nodules primarily on the face, although it can also affect the upper arms, trunk, and back. The pathogenesis of acne vulgaris involves the interaction of multiple factors that ultimately lead to the formation of its primary lesion, which is known as "comedo".

Because of its long duration and exposure to affected areas, acne is associated with a major deterioration in a patient's quality of life and well-being .

Up to 95% of acne sufferers have some degree of acne scarring, with 30% reporting severe acne scarring. Scarring from acne is common when medical care is delayed or is not sufficient, although it can also occur even when treatment is adequate .

About 90% of acne scars are related with collagen loss (atrophic scars), whereas the remaining 10- 20% show collagen gain (keloidal or hypertrophic scars). Resulting from the contraction of fibrous tissue, atrophic scars appear as depressions. Atrophic acne scars can be classified into three distinct types: boxcar, icepick, and rolling.

ELIGIBILITY:
Inclusion criteria:

patients aged equal or more than 18 years with atrophic post acne scars.

Exclusion criteria:

pregnancy and lactation. Hypertrophic scars. patients suffering from aggressive inflammatory acne. kidney or liver disease. active infection at site of lesion. patients use medications that reduce tissue healing during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of treating atrophic post acne scars with topical insulin versus PRP combined with fractional ablative Co2 laser. | 5 months from the beginning of the treatment
  Scar assessment will be made using the Goodman and Baron Qualitative and Quantitative scarring system at baseline and at each visit to evaluate the clinical improvement.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan HM, Zhao HJ, Guo DY, Zhu PQ, Zhang CL, Jiang W. Gut microbiota alterations in moderate to severe acne vulgaris patients. J Dermatol. 2018 Oct;45(10):1166-1171. doi: 10.1111/1346-8138.14586. Epub 2018 Aug 13. PMID 30101990
- [Background] Szepietowska M, Dabrowska A, Nowak B, Skinderowicz K, Wilczynski B, Krajewski PK, Jankowska-Konsur A. Facial acne causes stigmatization among adolescents: A cross-sectional study. J Cosmet Dermatol. 2022 Dec;21(12):6815-6821. doi: 10.1111/jocd.15268. Epub 2022 Oct 14. PMID 35869826
- [Background] Bhargava S, Cunha PR, Lee J, Kroumpouzos G. Acne Scarring Management: Systematic Review and Evaluation of the Evidence. Am J Clin Dermatol. 2018 Aug;19(4):459-477. doi: 10.1007/s40257-018-0358-5. PMID 29744784